CLINICAL TRIAL: NCT05466682
Title: RELAXaHEAD for Headache Patients (Phase II): RELAXaHEAD for Migraine and Sleep
Brief Title: RELAXaHEAD for Headache Patients (Phase II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Center for Advancing Point of Care Technologies (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00525-2
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Migraine; Headache; Multiple Sclerosis; Insomnia
Keywords: Progressive Muscle Relaxation Therapy; Migraine; Insomnia
MeSH Terms: conditions — Migraine Disorders; Headache; Multiple Sclerosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELAX (Experimental): Patients will receive Progressive Muscle Relaxation Therapy (PMR) via the RELAXaHEAD smart-phone app.
  Patients will be asked to do the following:
  * Week 1: 5 min deep breathing at least 5/7 days of the week
  * Week 2: 5 min PMR session at least 5/7 days of the week
  * Week 3: 15 min PMR session at least 5/7 days of the week
  * Week 4: PMR at least 4 days a week
  * Week 5: PMR at least 3 days a week
  * Weeks 6-8: Use PMR when it is most helpful
  Patients will be asked to track headache frequency, intensity, sleep, and acute medication use on the app. They will also receive written educational material about migraine.
  Interventions: Behavioral: Smartphone-Based Progressive Muscle Relaxation Therapy (PMR)
- Monitored Usual Care (MUC) (Active Comparator): Patients will be given a general education session consisting of basic migraine information. They will receive the RELAXaHEAD app but the Progressive Muscle Relaxation Therapy (PMR) function will be blocked.
  Patients will be asked to track headache frequency, intensity, sleep, and acute medication use on the RELAXaHEAD app. They will also receive written educational material about migraine.
  Interventions: Behavioral: Monitored Usual Care (MUC)

INTERVENTIONS:
Behavioral: Smartphone-Based Progressive Muscle Relaxation Therapy (PMR) — Relaxation technique delivered via RELAXaHEAD app.
  Arms: RELAX
Behavioral: Monitored Usual Care (MUC) — Standard of care plus daily symptom reporting using the RELAXaHEAD app electronic diary.
  Arms: Monitored Usual Care (MUC)

SUMMARY:
The goal of this research is to assess the utility of smartphone-based progressive muscle relaxation (PMR) for the treatment of migraine and sleep. While there are many commercially available electronic diary and mind-body intervention apps for headache, there is little data showing their efficacy. RELAXaHEAD app incorporates the electronic PMR that was successfully used in an earlier epilepsy study and beta tested with headache specialist and migraine patient input. It also is an electric headache diary. The app has been studied and findings have been reported in multiple peer reviewed publications. Also, the app has been updated based on prior feedback from the studies. Now, this 2-arm randomized controlled study will evaluate the feasibility and acceptability of RELAXaHEAD for use with patients with migraine and comorbid insomnia. . One arm will be the RELAX group (the RELAXaHEAD app) and the other arm will be a monitored usual care (MUC) group (this group receives standard of care and uses the electronic daily symptom reporting diary). The goals are to assess the feasibility and adherence of the RELAX intervention in persons with migraine and insomnia (Aim 1) and to gather exploratory data on the effects of the RELAX intervention on headache and sleep related outcome measures (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years (age 18-65 in urgent care);
* Meets migraine criteria based on the International Classification of Headache Disorders (ICHD) criteria;
* Migraine Disability Assessment (MIDAS) score >5. 4+ headache days a month OR; meets chronic post- traumatic headache (PTH) criteria based on International Classification of Headache Disorders (ICHD) criteria, is 3-12 months post-injury, and there are 4+ headache days a month.
* Scoring > or = 15 on the ISI.

Exclusion Criteria:

* Patients who have had Cognitive Behavioral Therapy, Biofeedback, or other Relaxation Therapy in the past year;
* Cognitive deficit or other physical problem with the potential to interfere with behavioral therapy;
* Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record;
* Opioid or barbiturate use 10+ days a month;
* Unable or unwilling to follow a treatment program that relies on written and audio file materials;
* Not having a smartphone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Dr. Minen (PI). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to alexis.george@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- RELAX: Patients will receive Progressive Muscle Relaxation Therapy (PMR) via the RELAXaHEAD smart-phone app.
  Patients will be asked to do the following:
  * Week 1: 5 min deep breathing at least 5/7 days of the week
  * Week 2: 5 min PMR session at least 5/7 days of the week
  * Week 3: 15 min PMR session at least 5/7 days of the week
  * Week 4: PMR at least 4 days a week
  * Week 5: PMR at least 3 days a week
  * Weeks 6-8: Use PMR when it is most helpful
  Patients will be asked to track headache frequency, intensity, sleep, and acute medication use on the app. They will also receive written educational material about migraine.
  Smartphone-Based Progressive Muscle Relaxation Therapy (PMR): Relaxation technique delivered via RELAXaHEAD app.
- Monitored Usual Care (MUC): Patients will be given a general education session consisting of basic migraine information. They will receive the RELAXaHEAD app but the Progressive Muscle Relaxation Therapy (PMR) function will be blocked.
  Patients will be asked to track headache frequency, intensity, sleep, and acute medication use on the RELAXaHEAD app. They will also receive written educational material about migraine.
  Monitored Usual Care (MUC): Standard of care plus daily symptom reporting using the RELAXaHEAD app electronic diary.
Period: Overall Study
Arm/Group | RELAX | Monitored Usual Care (MUC)
Started | 24 | 24
Completed | 22 | 21
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RELAX | Monitored Usual Care (MUC) | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Full Range); unit: years] | 43.5 [21 to 65] | 44.8 [26 to 69] | 44.2 [21 to 69]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Other | 0 | 1 | 1
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Enrolled in the Study
Description: Measure of feasibility.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 24 | 24
Participants | 24 | 24

2. Primary Outcome: Daily Diary Satisfaction Scores
Description: 5-item self-assessment measuring satisfaction with the daily dairy function of the RELAXaHEAD app. Items are ranked on a 5-point Likert scale, where: 0 = Strongly Disagree; 1 = Disagree; 2 = Neither Agree nor Disagree; 3 = Agree; and 4 = Strongly Agree.
  The total score is the sum of responses. Scores range from 0-20; higher scores indicate higher levels of satisfaction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 24 | 24
score on a scale | 4.2 (0.6) | 4.2 (0.3)

3. Primary Outcome: Daily Diary Satisfaction Scores
Description: as for outcome 2
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 23 | 23
score on a scale | 4.4 (0.6) | 4.2 (0.6)

4. Primary Outcome: Daily Diary Satisfaction Scores
Description: as for outcome 2
Time Frame: Month 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 18 | 19
score on a scale | 3.7 (1.1) | 3.4 (1.1)

5. Primary Outcome: Daily Diary Satisfaction Scores
Description: as for outcome 2
Time Frame: Month 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 17 | 20
score on a scale | 3.9 (0.9) | 3.4 (1)

6. Primary Outcome: Daily Diary Satisfaction Scores
Description: as for outcome 2
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 19 | 19
score on a scale | 3.6 (1.1) | 3.4 (0.9)

7. Primary Outcome: Progressive Muscle Relaxation Therapy (PMR) Satisfaction Scores Among RELAX Arm Participants
Description: 4-item self-assessment measuring satisfaction with PMR administered via the RELAXaHEAD app. Items are ranked on a 5-point Likert scale, where: 0 = Strongly Disagree; 1 = Disagree; 2 = Neither Agree nor Disagree; 3 = Agree; and 4 = Strongly Agree.
  The total score is the sum of responses. Scores range from 0-16; higher scores indicate higher levels of satisfaction
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX
Number analyzed (Participants) | 24
score on a scale | 3.7 (0.7)

8. Primary Outcome: Progressive Muscle Relaxation Therapy (PMR) Satisfaction Scores Among RELAX Arm Participants
Description: as for outcome 7
Time Frame: Week 1
Population: Monitored Usual Care (MUC) participants did not have data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX
Number analyzed (Participants) | 23
score on a scale | 4 (0.7)

9. Primary Outcome: Progressive Muscle Relaxation Therapy (PMR) Satisfaction Scores Among RELAX Arm Participants
Description: as for outcome 7
Time Frame: Month 1
Population: Monitored Usual Care (MUC) participants did not have data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX
Number analyzed (Participants) | 20
score on a scale | 3.5 (1.2)

10. Primary Outcome: Progressive Muscle Relaxation Therapy (PMR) Satisfaction Scores Among RELAX Arm Participants
Description: as for outcome 7
Time Frame: Month 2
Population: Monitored Usual Care (MUC) participants did not have data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX
Number analyzed (Participants) | 13
score on a scale | 3.5 (1.1)

11. Primary Outcome: Progressive Muscle Relaxation Therapy (PMR) Satisfaction Scores Among RELAX Arm Participants
Description: as for outcome 7
Time Frame: Month 3
Population: Monitored Usual Care (MUC) participants did not have data collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RELAX
Number analyzed (Participants) | 14
score on a scale | 3.9 (1.1)

12. Primary Outcome: Number of Days RELAX Arm Participants Performed Progressive Muscle Relaxation Therapy (PMR) at Least 5 Minutes/Day
Description: Calculated using the backend analytics in the RELAXaHEAD app. Measure of feasibility.
Time Frame: Up to Month 3
Population: Monitored Usual Care (MUC) participants did not have data collected.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RELAX
Number analyzed (Participants) | 19
Days | 22.1 (27.6)

13. Primary Outcome: Number of Days Participants Used Diary
Description: Calculated using the backend analytics in the RELAXaHEAD app. Measure of feasibility.
Time Frame: Up to Month 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RELAX | Monitored Usual Care (MUC)
Number analyzed (Participants) | 24 | 24
Days | 54.58 (31.88) | 62.08 (27.27)

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-cause mortality was not assessed in the study population.
Arm/Group | RELAX | Monitored Usual Care (MUC)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT05466682/Prot_SAP_000.pdf